CLINICAL TRIAL: NCT03600207
Title: The Effect of Diaphragm Muscle Training on Chronic Low Back Pain
Acronym: LBP_DT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Szeged University (Other)
Responsible Party: Principal Investigator, Tamás Bender, Clinical Professor, Szeged University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LBP_DT_001
Record Dates: First submitted 2018-06-21; First posted 2018-07-26 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Low Back Pain; Diaphragm
Keywords: Low Back Pain; Diaphragm
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group -complex training (Active Comparator): complex training
  Interventions: Other: Complex training
- Experimental group -diaphragm training (Active Comparator): diaphragm training
  Interventions: Other: Complex training; Other: Diaphragm training

INTERVENTIONS:
Other: Complex training — The training program contains stretching, mobilizing, strengthening exercises on the trunk and hip muscles and a proprioceptive training.
Other: Diaphragm training — The training program contains strengthening exercises on the diaphragm muscle.
  Arms: Experimental group -diaphragm training

SUMMARY:
Brief Summary: Low back pain is very common problem in all the developed countries and affects children to elderly. Based on the etiology the low back pain is divided into two type: nonspecific and specific low back pain. If the pathological reason is known it is defined as specific and if the reason for the pain is unknown it is defined as nonspecific low back pain. The postulated reason for nonspecific low back pain is the segmental instability of the lumbar spine. Diaphragm muscle has a role in maintaining the segmental stability. The aim of this study to reduce the severity of the low back pain with improving the stability of the lumbar spine by using diaphragm training.

DETAILED DESCRIPTION:
The study is a randomized controlled trial. The participants are divided randomly into two groups. One of the groups take part in a complex training which contains stretching, strengthening, mobilizing exercises and proprioceptive training and this training is completed by diaphragm strengthening exercises. This group is defined as diaphragm training group. The members of the diaphragm training group use the POWERbreathe Medic Plus device. Opposed to the diaphragm training group the members of the control group take part only in the complex training without strengthening the diaphragm muscle. The pain intensity is assessed by Visual Analogue Scale and the diameter of the stabilizer muscles' belly is measured by B-mode ultrasound examination, using Zonare Z.One Ultrasound System (Mountain View, CA, USA). The thickness of the transversus abdominis muscle, the lumbar multifidus muscle and the diaphragm muscle is assessed in two different positions: during lying and during sitting position with weightlifting. The muscles are measured in two different states: a relaxed and a contracted state. Functional tests and a balance platform (NeuroCom) are used to measure the stability, and the function of the diaphragm is assessed by using a POWERbreathe KH2 device.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain
* Do not take part in other treatment
* Be able to learn the usage of diaphragm trainer

Exclusion Criteria:

* Balance problems with neurological cause
* Malignant tumor
* Serious organ disease
* Respiratory disease
* A previous surgical intervention which affected the trunk
* The patient is unable to cooperate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Pain assessed by Visual Analogue Scale (followed by its scale information in the Description) | 8 weeks
  The severity of the pain is measured with Visual Analogue Scale (VAS) before and after the intervention. This is a semi-objective, self-report device that is used extensively to measure such complaints as pain. The sclale is a 10 cm line. The scale is anchored by 'no pain' (0 score) and 'worst imaginable pain' (score of 10). Therefore the higher values represent a worse outcome. When using the Visual Analogue Scale, the participants had to mark on a 10 cm long line the average severity of lumbar pain and we measured the distance of their mark from the zero point in cm-s.
Thickness of the stabilizer muscles' belly | 8 weeks
  The thickness of the stabilizer muscles's belly is measured with an ultrasound examination (Zonare Z.One Ultrasound System). The assessed muscles are transversus abdominis muscle, diaphragm muscle and lumbar multifidus muscle before and after the intervention.

SECONDARY OUTCOMES:
Respiratory muscles' function | 8 weeks
  Respiratory muscles' function is measured with POWERbreathe KH2 device before and after the intervention.
Limits of stability in sitting | 8 weeks
  It is measured by modified Functional and Lateral Reach Test before and after the intervention. Modified means the sitting position.
Functional skills | 8 week
  The functional skills are measured by the standard Timed Up and Go Test, Four Square Step Test and Fingertip to Toe Test before and after the intervention.
Balance and stability | 8 weeks
  The balance and the stability of the participants is measured with a force platform (NeuroCom Basic Balance Master) using CTSIB and Unilateral Stance protocol before and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- SZTE-Egészségtudományi és Szociális Képzési Kar, Szeged, Hungary